CLINICAL TRIAL: NCT05653401
Title: Treatment of Renal Colic in the Emergency Department: Comparison Between Magnesium Sulfate and Lidocaine. A Double-blind, Randomised Controlled Trial.
Brief Title: Treatment of Renal Colic in the Emergency Department: Comparison Between Magnesium Sulfate and Lidocaine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMonastir2022
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Renal Colic
Keywords: Acute pain; Renal colic; Magnesium Sulfate; Lidocain; Diclofenac
MeSH Terms: conditions — Renal Colic; Acute Pain | interventions — Magnesium Sulfate; Diclofenac

STUDY DESIGN:
Intervention Model Description: Double blind study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium Sulfate (Active Comparator): Intravenous Magnesium Sulfate combined to Diclofenac
  Interventions: Drug: Magnesium sulfate and diclofenac
- Lidocaine (Active Comparator): Intravenous lidocaine combined to Diclofenac
  Interventions: Drug: Lidocain and diclofenac
- Diclofenac (Active Comparator): Intramuscular Diclofenac alone
  Interventions: Drug: Placebo and diclofenac

INTERVENTIONS:
Drug: Magnesium sulfate and diclofenac — Intramuscular injection of 75 mg/ 3 ml of Diclofenac solution Intravenous injection of 1 g of Magnesium Sulfate solution diluted in 10 ml of saline solution administered over 2 to 4 minutes
  Other Names: Intravenous Magnesium Sulfate combined to Diclofenac
  Arms: Magnesium Sulfate
Drug: Lidocain and diclofenac — Intramuscular injection of 75 mg/ 3 ml of Diclofenac solution Intravenous injection of 10 ml of Lidocaine 1% solution administered over 2 to 4 minutes.
  Other Names: Intravenous Lidocain combined to Diclofenac
  Arms: Lidocaine
Drug: Placebo and diclofenac — Intramuscular injection of 75 mg of Diclofenac solution and 10 ml Intravenous injection of serum saline ( as a Placebo Comparator ) administered over 2 to 4 minutes.
  Other Names: Diclofenac alone with placebo ( serum saline )
  Arms: Diclofenac

SUMMARY:
Rate of Intravenous Magnesium Sulfate Vs Lidocaine to treat Renal Colic in the Emergency Department.

DETAILED DESCRIPTION:
Magnesium Sulfate (MgSO4) is a N-Methyl-D-aspartate (NMDA) receptor antagonist and is thought to be involved in the modulation of pain. There has been little direct evidence that MgSO4 relieve neuropathic pain and prevents opioid-induced hyperalgesia in humans.

Intramuscular Diclofenac seems to offer the most effective sustained analgesia for renal colic in the ED and has few side effects.

Lidocain became the agent of choice in visceral and central pain. Intravenous Lidocain is effective in the management of neuropathic pain such as diabetic neuropathy, post-surgical pain, post-herpetic pain, headaches and neurological malignancies. At low doses, Lidocain is known as a relatively safe medication. Lidocain seems an effective treatment who can be administrated in the renal colic.

Objective of study:

Evaluate the analgesic effect of a standard dose of intravenous magnesium added to intramuscular diclofenac compared to intravenous Lidocain combined to intramuscular diclofenac or intramuscular diclofenac alone in patients presenting to the ED with renal colic and whether it can reduce opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Age between 18 and 65 years .
* Diagnosis of renal colic made by an emergency medicine physician, based on history and clinical findings, and urine analysis or by identifying the urinary tract stone using ultrasonography or radiologic imaging including CT scan .-With moderate to severe pain (visual analogic Scale ≥5 ).

Exclusion Criteria:

* known renal or hepatic dysfunction, use of NSAIDs and/or opioids within 6 h before presentation
* history of bleeding diathesis, history of peptic ulcer disease or gastrointestinal hemorrhage,
* History of cardiac arrhythmia, severe coronary artery disease, seizures, presence of any peritoneal sign, altered mental status, and anticoagulant medication or coagulation disorders.
* Use of any analgesics or spasmolytics in the previous 4 hours before admission, hemodynamic instability, and prior known allergy to lidocaine or morphine .
* Pregnant women , Breast feeding
* Allergy or contraindications to NSAIDs, lidocaine or MgSO 4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment success evaluated By VAS Score ( 10 cm Visual analogue Score ) 30 minutes after drug administration. | 30 minutes
  Significant pain reduction as at least a 50% drop of VAS Score of the initial pain score at 30 min after analgesia administration ( Drop VAS Score is in favour of analgesic treatment efficiency )

SECONDARY OUTCOMES:
The proportion of participants with persistent pain (VAS > 2) at the end of the study (90 min) | 90 min
  The proportion of participants with persistent pain (VAS > 2) at the end of the study (90 min)
Adverse effect | 90 minutes
  nausea, vomiting, vertigo, and lethargy based on self-reports and other clinical manifestations occuring at any moment of the protocol
The need for additional analgesics at 30 minutes after protocol start to relieve the pain | 30 minutes
  The need for rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No